CLINICAL TRIAL: NCT02447588
Title: Programming IUI With Sperm Donor in Patients With High Progesterone the Day of hCG Administration
Brief Title: IUI Schedule in Cases of High Progesterone
Acronym: IAD-P4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IVI Madrid (Other)
Collaborators: Vida Recoletas Sevilla (Other); IVI Vigo (Other)
Responsible Party: Principal Investigator, Antonio Requena, PhD MD, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1504-MAD-021-AR
Record Dates: First submitted 2015-05-07; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Infertility
Keywords: intrauterine insemination; progesterone
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Intrauterine insemination with sperm donor (IAD) at 36 hours post-hCG. Cases where the IAD is scheduled at 36 hours post-administration of hCG.
  Interventions: Other: IAD at 36 hours
- Group 2 (Experimental): Intrauterine insemination with sperm donor (IAD) at 24 hours post-hCG. Cases where the IAD is scheduled at 24 hours post-administration of hCG.
  Interventions: Other: IAD at 24 hours

INTERVENTIONS:
Other: IAD at 36 hours — Intrauterine insemination with sperm donor at 36 hours post-hCG
  Arms: Group 1
Other: IAD at 24 hours — Intrauterine insemination with sperm donor at 24 hours post-hCG
  Arms: Group 2

SUMMARY:
Intrauterine insemination (IUI) combined with ovarian stimulation protocols has become one of the first alternative treatment against infertility, although results in gestational terms are highly variable, ranging between 10% and 25%. The influence of progesterone levels in stimulated cycles of intrauterine insemination is an aspect little studied; however, this information may be useful when synchronizing the time of insemination with the implantation window, as it has been observed that patients with elevated levels of progesterone in the follicular phase exhibit a significant decrease in ongoing pregnancy rates, these results being possible due to premature ovulation which causes asynchrony between the embryo and the endometrium.

Taking into account these considerations, the aim of the investigators' study is to determine the effectiveness, in terms of ongoing pregnancy rates, to advance the intrauterine insemination with sperm donor (24 hours post-hCG) with respect to the standard schedule (36 hours post-hCG) according progesterone levels determined the day of hCG administration

DETAILED DESCRIPTION:
Correct schedule of intrauterine insemination is essential to the success of these treatments due to the limited range in which the capacitated sperm survive the female genital tract and oocytes can be fertilized after ovulation. For intrauterine insemination, the fraction of motile sperm is injected directly into the uterine cavity and later migrate into abdominal cavity, where they remain a few hours after insemination; meanwhile, fertilizable oocytes are only between 12-16 hours after ovulation. In the cycles in which follicular growth is monitored, a spontaneous LH surge before ovulation induction with HCG is a possibility; indeed, in stimulated cycles LH is not usually determined so clinicians are not able to know if there has been or not ovulation. Ovulation usually occurs 24 hours after the LH surge; therefore, an insemination performed 36 hours after ovulation induction may be too late in cases of premature ovulation.

The influence of progesterone levels in stimulated cycles of intrauterine insemination is an aspect little studied; however, this information can be useful when synchronizing the time of insemination with the implantation window.

The day of ovulation induction, the investigators will determine progesterone levels. If progesterone> 1 ng / ml the patient be randomized in one of the following groups:

* Group 1 (intrauterine insemination with sperm donor IAD at 36 hours post-hCG). Cases where the IAD is scheduled at 36 hours post-administration of hCG.
* Group 2 (IAD at 24 hours post-hCG). Cases where the IAD is scheduled at 24 hours post-administration of hCG.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18-30 kg / m2
* Patent tubes
* Regular cycles (26-35 days)
* FSH levels on day 3 of cycle (<10 mIU / ml)
* Estradiol levels on day 3 of cycle (<60 pg / ml)
* Progesterone levels the day of hCG (> 1 ng / ml)
* Semen donors belonging to the bank of IVI

Exclusion criteria

* Patients with ≥3 follicles of over 16 mm diameter
* No dominant follicle after two consecutive ultrasound
* Women with P <1 ng / ml on the day of hCG

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 1 month

SECONDARY OUTCOMES:
Doses of gonadotropins | 1 day
Estradiol levels the day of hCG administration | 1 day
LH levels the day of hCG administration | 1 day
Days of stimulation | 1 day
Cancellation rate | 1 month
Pregnancy rate | 1 month
Miscarriage rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Requena, PhD, MD, Principal Investigator — IVI Madrid

REFERENCES:
- [Background] Venetis CA, Kolibianakis EM, Papanikolaou E, Bontis J, Devroey P, Tarlatzis BC. Is progesterone elevation on the day of human chorionic gonadotrophin administration associated with the probability of pregnancy in in vitro fertilization? A systematic review and meta-analysis. Hum Reprod Update. 2007 Jul-Aug;13(4):343-55. doi: 10.1093/humupd/dmm007. Epub 2007 Apr 3. PMID 17405832
- [Result] Antaki R, Dean NL, Lapensee L, Racicot MH, Menard S, Kadoch IJ. An algorithm combining ultrasound monitoring and urinary luteinizing hormone testing: a novel approach for intrauterine insemination timing. J Obstet Gynaecol Can. 2011 Dec;33(12):1248-52. doi: 10.1016/s1701-2163(16)35110-6. PMID 22166279
- [Result] Azem F, Tal G, Lessing JB, Malcov M, Ben-Yosef D, Almog B, Amit A. Does high serum progesterone level on the day of human chorionic gonadotropin administration affect pregnancy rate after intracytoplasmic sperm injection and embryo transfer? Gynecol Endocrinol. 2008 Jul;24(7):368-72. doi: 10.1080/09513590802196353. PMID 18645708
- [Result] Blockeel C, Knez J, Polyzos NP, De Vos M, Camus M, Tournaye H. Should an intrauterine insemination with donor semen be performed 1 or 2 days after the spontaneous LH rise? A prospective RCT. Hum Reprod. 2014 Apr;29(4):697-703. doi: 10.1093/humrep/deu022. Epub 2014 Feb 18. PMID 24549212